CLINICAL TRIAL: NCT04705974
Title: Minimum Effective Dose of Ropivacaine for Peripheral Nerve Block on Posture-evoked Pain for Spinal Anesthesia in Patients With Hip Fracture
Brief Title: MED90 of Ropivacaine for Peripheral Nerve Block on Posture-evoked Pain in Spinal Anesthesia Positioning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: MEDNB-HP
Record Dates: First submitted 2021-01-09; First posted 2021-01-12 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fascia iliaca block (Experimental): ultrasound-guided fascia iliaca block with predetermined dose of 0.4% ropivacaine will be performed.
  Interventions: Procedure: Fascia iliaca block
- Femoral nerve block (Experimental): ultrasound-guided ultrasound-guided femoral nerve block with predetermined dose of 0.4% ropivacaine will be performed.
  Interventions: Procedure: Femoral nerve block
- Pericapsular nerve group block (PENG block) (Experimental): ultrasound-guided ultrasound-guided pericapsular nerve group block with predetermined dose of 0.4% ropivacaine will be performed.
  Interventions: Procedure: Pericapsular nerve group block (PENG block)

INTERVENTIONS:
Procedure: Fascia iliaca block — Fascia iliaca block will be performed under ultrasound guidenance.
  Arms: Fascia iliaca block
Procedure: Femoral nerve block — Femoral nerve block will be performed under ultrasound guidenance.
  Arms: Femoral nerve block
Procedure: Pericapsular nerve group block (PENG block) — Pericapsular nerve group block (PENG block) will be performed under ultrasound guidenance.
  Arms: Pericapsular nerve group block (PENG block)

SUMMARY:
This study aims to determine the minimum effective dose of ropivacaine for peripheral nerve block on posture-evoked pain for spinal anesthesia in elderly patients with hip fracture. Three types of peripheral nerve block, including fascia iliaca block, femoral nerve block and Pericapsular nerve group block (PENG block) will be assessed.

DETAILED DESCRIPTION:
Patients with hip fractures are anticipated to endure sever pain caused by positional changes required for spinal anesthesia. Providing analgesia before positioning not only increases patient comfort but also improves positioning and successful spinal block. Peripheral nerve block is an effective strategy for relieving pain during postures change for spinal anesthesia in patients with hip fractures. Three types of peripheral nerve block, including fascia iliaca block, femoral nerve block and Pericapsular nerve group block (PENG block), has been successfully used for analgesia for spinal anesthesia positioning in patients with hip fractures. However, the minimum effective dose of local anesthetics for these three types of peripheral nerve block is not known. This study aims to determine the minimum effective dose of ropovacaine in the three types of peripheral nerve block using a biased coin design up-and-down sequential method. Successful block is defined as NRS score ≤3 by positional changes for spinal anesthesia, achieved at 20min after the block. MED90 of ropivacaine for fascia iliaca block, femoral nerve block and PENG block be assessed respectively. Patients will receive ultrasound guided peripheral nerve block. The initial dose is chosen as 80 mg on the basis of clinical experience. Subsequently, if a patient has an inadequate block, the ropivacaine dose is increased by 8 mg in the next subject. If a patient has a successful block, the next subject is randomized to receive either a lower dose (with a decrement of 8 mg), with a probability of b = 0.11, or the same dose, with a probability of 1 - b = 0.89. Forty five successful blocks for each type of nerve block will be accomplished. MED90 of each type of nerve block will be calculated by isotonic regression.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 - 85 years
* American Society of Anesthesiologists physical statusⅠ- Ⅲ
* Patients will receive hip replacement

Exclusion Criteria:

* Patient refusal
* Cognitive impairment(NRS pain score cannot be assessed)
* Peripheral neuropathy
* Mutiple furacture
* skin infection at the site of injection
* allergy to ropivacaine、lidocaine or bupivacaine
* contraindication to spinal anesthesia

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
The minimum effective dose of ropivacaine in three types of nerve block for analgesia for spinal anesthesia positioning in patients with hip fractures | up to 24 months
  The minimum effective dose of ropivacaine in each type of nerve block is based on 45 patients with satisfactory analgesia during positioning for spinal anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No